CLINICAL TRIAL: NCT01401595
Title: Brain Imaging and Treatment Studies of the Night Eating Syndrome
Acronym: NES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Kelly Allison, Assistant Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 806753
Record Dates: First submitted 2011-05-23; First posted 2011-07-25 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Night Eating Syndrome
MeSH Terms: conditions — Night Eating Syndrome | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Night Eaters (Experimental): Subjects will be given a medical history, height and weight will be measured, and BMI calculated. Initial outpatient assessment will include diary measurement of food intake and nighttime awakenings (and associated food intake) together with psychological testing. For women, a pregnancy test will also be administered no more than 48 hours before SPECT-CT imaging and the beginning of escitalopram oxalate (Lexapro) treatment. Escitalopram oxalate (Lexapro) open-label treatment will last 12 weeks. Dosing will start at 10 mg and increase to 20 mg per day flexibly. Treatment will be discontinued starting at 12 weeks under the supervision of our study physician.
  Interventions: Drug: escitalopram oxalate
- Control Subjects (No Intervention): At the beginning of the study, control subjects will be given a medical history, height and weight will be measured, and BMI calculated. Initial outpatient assessment will include diary measurement of food intake and nighttime awakenings (and associated food intake) together with psychological testing.
  An ADAM SPECT or SPECT-CT study of SERT binding will be conducted which will compare SERT binding of the 10 control subjects with that of the 30 night eating subjects. The first procedure will be to assess SPECT or SPECT-CT images of night eaters and controls following up our pilot SPECT study of night eaters and controls.

INTERVENTIONS:
Drug: escitalopram oxalate — The purpose of this study is to determine the effectiveness of the anti-depressant Lexapro in the treatment of the Night Eating Syndrome. An ADAM SPECT-CT study of SERT binding will be conducted which will compare SERT binding in 31 night eaters with that of 10 control subjects. The first procedure will be to assess SPECT-CT images of night eaters and controls following up our pilot SPECT study of night eaters and controls. Medication will be administered starting at 10 mg daily, with increase up to 20 mg, as indicated and tolerated, for up to three months. Visits will occur at baseline and weeks 1, 2, 4, 6, 8, 10, and 12.
  Other Names: Lexapro
  Arms: Night Eaters

SUMMARY:
The purpose of this study is to determine the effectiveness of the anti-depressant Lexapro in the treatment of the Night Eating Syndrome.

DETAILED DESCRIPTION:
This proposal explores the implications of our two recent major discoveries: the striking efficacy of the Selective Serotonin Reuptake Inhibitor (SSRI) sertraline in the control of the Night Eating Syndrome (NES) and the unprecedented elevation in the level of serotonin transporter (SERT) binding in the midbrain of persons with NES. Our overall theory is that NES is associated with a syndrome-specific increase in SERT derived from a genetic vulnerability which is affected by life stress. This increased SERT activity produces a fall in post-synaptic serotonin levels. The investigators hypothesize that these decreased serotonin levels result in a significant phase delay in circadian food intake manifested by evening hyperphagia, nighttime ingestions and morning anorexia. SSRIs that block this increased SERT activity increase synaptic serotonin levels and restore the circadian rhythm of food intake.

ELIGIBILITY:
Inclusion Criteria:

* men and women suffering from NES
* ages 18 to 70 years
* BMI greater than 18.5 kg/m2

Exclusion Criteria:

* Children or adolescents <18 years
* persons older than 70
* patients with diabetes mellitus
* thyroid disease and other endocrine and metabolic disorders
* use within the past month of any psychotropic medication, oral steroids, diuretics or hypnotics
* current anorexia nervosa or bulimia nervosa
* participation in an organized weight reduction program
* use of antiobesity medication
* an occupation that involves night shifts or other unusual time requirements -Major Depressive Disorder (judged severe)
* Bipolar Disorder
* suicidal risk
* current or past psychosis
* substance use or abuse disorder within the past 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C Allison, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- The Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Allison KC, Studt SK, Berkowitz RI, Hesson LA, Moore RH, Dubroff JG, Newberg A, Stunkard AJ. An open-label efficacy trial of escitalopram for night eating syndrome. Eat Behav. 2013 Apr;14(2):199-203. doi: 10.1016/j.eatbeh.2013.02.001. Epub 2013 Mar 5. PMID 23557820
- See also: The Center for Weight and Eating Disorders — http://www.med.upenn.edu/weight/research.shtml

RESULTS

PARTICIPANT FLOW:
Groups:
- Night Eaters: Subjects were given a medical history, and height and weight was measured. Initial outpatient assessment included diary measurement of food intake and nighttime awakenings (and associated food intake) together with psychological testing. For women, a pregnancy test was also administered no more than 48 hours before SPECT-CT imaging and the beginning of Lexapro treatment. Lexapro treatment lasted 12 weeks.
  escitalopram oxalate: The purpose of this study is to determine the effectiveness of the anti-depressant Lexapro in the treatment of the Night Eating Syndrome. An ADAM SPECT-CT study of SERT binding was conducted which will compare SERT binding in 30 night eaters with that of 10 controls. The first procedure assessed SPECT-CT images of night eaters and controls. Medication was administered starting at 10 mg daily, with increases up to 20 mg, as indicated and tolerated, for up to three months. Visits occured at baseline and weeks 1, 2, 4, 6, 8, 10, and 12.
- Control Subjects: At the beginning of the study, control subjects were given a medical history, height and weight was measured, and BMI calculated. Initial outpatient assessment included diary measurement of food intake and nighttime awakenings (and associated food intake) together with psychological testing.
  An ADAM SPECT-CT study of SERT binding was conducted which will compare SERT binding of the 10 control subjects with that of the 30 night eating subjects to assess SPECT-CT images of night eaters and controls following up our pilot SPECT study of night eaters and controls.
Period: Recruitment and Screening
Arm/Group | Night Eaters | Control Subjects
Started | 75 (Of 345 calls, 75 potential NES subjects attended the screening visit and provided informed consent.) | 12 (Of 32 calls, 12 control subjects attended an initial screening visit.)
Completed | 32 (Of the 75, 32 remained interested/eligible after the initial screening period.) | 10 (10 of the 12 remained eligible/interested after the initial screening visit.)
Not Completed | 43 | 2
Period: Imaging and Treatment (for NE Arm)
Arm/Group | Night Eaters | Control Subjects
Started | 32 | 10
Completed | 18 | 10
Not Completed | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Night Eaters: 31 participants screened and diagnosed with NES attended the baseline treatment session and at least one follow-up appointment.
- Control Subjects: 10 control participants completed the baseline screening and SPECT scans.
- Total: Total of all reporting groups
Arm/Group | Night Eaters | Control Subjects | Total
Number analyzed (Participants) | 31 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 10 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 6 | 27
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 29 | 7 | 36
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 4 | 16
  White | 15 | 4 | 19
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms of NES
Description: Outcome of treatment will be measured by self report questionnaire, the Night Eating Symptom Scale ( higher score indicates worse symptoms). The percentage of calories consumed after dinner was estimated by recall at each treatment visit, as compared to their baseline % of intake after dinner, which was calculated through food diaries. The number of nocturnal ingestions (waking during the night and eating) per week was also recalled at each treatment visit.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percentage of calories after dinner
Groups:
- Night Eating Syndrome Open Label Escitalopram Treatment: All subjects with NES participated in the open label treatment with escitalopram, although of the 32 participants, 1 did not return after her initial medication visit. As it is unknown if this participants started the medication, only the 31 participants who returned to a second visit or more were included in the analysis
- Controls: The control participants did not participate in the treatment part of the study - only the baseline SPECT scans.
Arm/Group | Night Eating Syndrome Open Label Escitalopram Treatment | Controls
Number analyzed (Participants) | 31 | 10
percentage of calories after dinner
  baseline %calories consumed after dinner | 46.1 (3.0) | 11.8 (2.4)
  treatment end %calories after dinner | 17.4 (3.5) | NA (NA) — Controls did not participate in the escitalopram treatment.

2. Secondary Outcome: Nocturnal Ingestions
Description: Number of nocturnal ingestions (waking and having something to eat) were reported at each visit.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Night Eating Syndrome Open Label Escitalopram Treatment: All NES subjects received the open label escitalopram treatment
- Controls: The controls did not participate in the escitalopram treatment portion of the study. The just completed the baseline screening and SPECT scan.
Arm/Group | Night Eating Syndrome Open Label Escitalopram Treatment | Controls
Number analyzed (Participants) | 31 | 10
units on a scale
  baseline nocturnal ingestions/week | 5.8 (0.5) | 0.0 (0.0)
  treatment end nocturnal ingestions/week | 1.2 (0.6) | NA (NA) — Controls did not participate in the escitalopram treatment.

3. Secondary Outcome: Night Eating Symptoms
Description: The responses on the Night Eating Symptom Scale (NESS) will be examined over time.
  Subjects will complete the NESS at their baseline visit, and at every treatment visit thereafter. The Night Eating Symptom Scale-II (NESS-II) (Lundgren, Allison, Vinai, & Gluck, 2012) is a 14-item questionnaire (possible range of 0-56, with higher scores indicating more severe symptoms) that assesses the presence of NES features over the course of the previous week. The NESS will indicate whether or not escitalopram is having an effect on our participants' night eating symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Night Eating Syndrome Open Label Escitalopram Treatment | Controls
Number analyzed (Participants) | 31 | 10
units on a scale
  Baseline Night Eating Symptom Scale | 30.2 (1.3) | NA (NA) — The NESS was administered at the first treatment visit, not at the baseline screening/characterization visit, so the controls did not complete this measure.
  treatment end night eating symptom scale | 15.2 (1.5) | NA (NA) — The controls did not participate in the escitalopram treatment.

ADVERSE EVENTS:
Time Frame: Duration of the study - 12 weeks, open label with escitalopram oxalate
Groups:
- Night Eating Syndrome Open Label Treatment Group: Only the 32 participants with NES participated in the open label escitalopram treatment trial. One participant did not return after the first visit, and it is unknown if she ever started the medication. Thus 31 participants were included in the statistical analyses.
Arm/Group | Night Eating Syndrome Open Label Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 5/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Night Eating Syndrome Open Label Treatment Group (N=31)
nausea (Gastrointestinal disorders) | 5
drowsiness (Nervous system disorders) | 4
dry mouth (General disorders) | 3
increased sweating (General disorders) | 2
impotence/low libido (Reproductive system and breast disorders) | 2
headache (Nervous system disorders) | 2
mental cloudiness (Nervous system disorders) | 2
diarrhea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No